CLINICAL TRIAL: NCT00001406
Title: Eosinophil Activation and Function in Parasitic Infections and Other Conditions With Increased Tissue or Peripheral Blood Eosinophilia in Humans
Brief Title: Activation and Function of Eosinophils in Conditions With Blood or Tissue Eosinophilia
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940079; 94-I-0079
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-02-28

CONDITIONS: Immune System Diseases; Eosinophilia; Helminthiasis; Hypersensitivity; Parasitic Disease
Keywords: Eosinophils; Helminth Parasites; Hypereosinophilia; Allergy; Asthma; Natural History
MeSH Terms: conditions — Immune System Diseases; Eosinophilia; Helminthiasis; Hypersensitivity; Parasitic Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Volunteers with elevated eosinophil counts in the peripheral blood or tissues; or a relative of a volunteer with eosinophilia

SUMMARY:
This study will investigate how, why and under what conditions eosinophils (a type of white blood cell) become activated and will examine their function in immune reactions. Eosinophil counts often rise in response to allergies, asthma, and parasitic worm infections. They can also go up in uncommon autoimmune conditions and, rarely, in association with tumors. Elevated levels of these cells is called eosinophilia. Usually, eosinophilia causes no apparent symptoms, but in rare cases there may be local swelling and itching, allergic lung problems, heart disease or nerve damage caused by the release of toxic substances in these cells into body tissues.

Patients 1 to 100 years of age with eosinophil counts greater than 750/ml or an abnormal accumulation of eosinophils in the skin or body tissues may be eligible for this study. All participants will have a thorough medical history, physical examination and blood tests. Depending on the person's age and symptoms, other diagnostic tests may be done, including specialized studies of the eye, lungs, skin, bone marrow, nerves or heart. This is not a treatment study, and no experimental treatments will be offered. Patients who require treatment will receive standard medical care.

Certain other procedures may be requested solely for research purposes. All participants will be asked to donate extra blood for laboratory studies investigating how immune cells and other immune substances in the blood act to stimulate a rise in eosinophils. In addition, some participants may undergo one or more of the following:

* Annual Follow-up evaluations - Physical examinations and blood tests to evaluate changes in the patient's condition and eosinophil counts over time.
* Bone marrow biopsy and aspiration will be recommended during the initial evaluation, and in certain patients at other times when it is important to look directly at the newly developing cells in the bone marrow. For this procedure an area of skin and bone is anesthetized with xylocaine (an anesthetic similar to that used by dentists), and a very sharp needle is used to sample the bone marrow for evaluation. Bone marrow biopsy and aspiration can have side effects of pain and/or bleeding into the skin and soft tissues at the site of the procedure. Rarely the area at the biopsy site can become infected, and is treated with antibiotics.
* Genetic testing: Some of the blood drawn from you as part of this study will be used for genetic tests. Genetic tests can help researchers study how health or illness is passed on to you by your parents or from you to your children. Any genetic information collected or discovered about you or your family will be confidential.
* Leukapheresis (only patients 18 years and older) to collect large numbers of certain cells - In this procedure, whole blood is collected through a needle placed in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are then removed and the rest of the blood is returned to the body, either through the same needle used to draw the blood or through a second needle placed in the other arm.

DETAILED DESCRIPTION:
Study Description: This study is designed to collect data and clinical samples from participants with elevated eosinophil counts in the peripheral blood or tissues or their relatives to enhance our understanding of the mechanisms driving eosinophilia and eosinophil activation in patients with a wide range of eosinophilic disorders with the ultimate goal of improving diagnostics and identifying novel treatment modalities for these patients. Eosinophilic participants will undergo an extensive clinical evaluation at baseline and at least yearly thereafter focused on the identification of the cause of eosinophilia and the presence of end organ manifestations. Blood, bone marrow, tissue, and/or body fluids will be collected for research purposes at initial and follow-up visits to address broader questions relating to the varied etiologies of eosinophilia, biomarkers of disease activity and eosinophil activation, and the functional role of eosinophils in homeostasis and disease pathogenesis. While this protocol is not primarily designed to study treatment of eosinophilic patients, the clinical and immunological responses to therapy will be monitored. This protocol will also allow clinical and laboratory evaluation of family members of subjects with eosinophilia to help identify genetic causes of eosinophilia and to provide controls for immunologic studies.

Objectives:

Primary Objective: to understand the mechanisms driving eosinophilia and eosinophil activation in patients with a wide range of eosinophilic disorders

Secondary Objectives:

1. To develop a diagnostic algorithm that accurately classifies eosinophilic patients by underlying etiology
2. To determine the mechanisms underlying eosinophil activation and recruitment to the blood and tissues
3. To understand the mechanisms of action of therapeutic agents used or in development for the treatment of HES
4. To assess the signs and symptoms experienced by patients with HES

Exploratory Objectives:

1. To investigate the multifunctional role of eosinophils in settings other than HES
2. To understand the long-term effects of eosinophilia in patients with HES
3. To assess the effects of race, sex, ethnicity, and environmental factors on the prevalence and clinical manifestations of eosinophilic disorders

Endpoints:

Primary Endpoint:

Identification and characterization of clinical and genetic variants of hypereosinophilic syndromes (HES)

Secondary Endpoints:

1. Identification of laboratory and clinical tests that distinguish between clinical and genetic variants of HES

2a. Identification of biomarkers of disease activity and specific organ involvement in eosinophilic disorders

2b. Identification of new therapeutic targets for the treatment of HES

3. Delineation of the effects of therapeutic agents on eosinophil development, activation, recruitment to tissues and/or apoptosis

4. Creation of a patient-related outcomes questionnaire for use in future treatment studies of HES

Exploratory Endpoints:

1. Description of the consequences of eosinophilia and/or eosinophil depletion in the context of varied immunologic and inflammatory

   settings
2. Collection of standardized longitudinal data on disease activity and outcome in patients with hypereosinophilia.
3. Comparison of prevalence and clinical manifestations of eosinophilic disorders among varied subpopulations of patients

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged 1-100
3. Ability of subject (or Legally Authorized Representative (LAR)) to understand and sign a written informed consent document

   Eosinophilic Patients only:
4. Documented peripheral blood count >1500/mm3, tissue eosinophilia (abnormal accumulation of eosinophils in the skin or other body tissues) or suspected eosinophilic end organ involvement
5. Primary (non-NIH) physician for routine medical care

   Relatives only:
6. Extended family member of an eosinophilic participant on this protocol

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any condition(s) or diagnosis, physical and/or psychological, that the investigator feels precludes the patient from participation in the study.

   Relatives only:
2. Females must not be pregnant

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with marked eosinophilia, eosinophilia in tissues or suspected eosinophilic end organ involvement will be seen on this protocol. Evaluation of family members may be of interest when a genetic cause of eosinophilia in suspected in a study participant.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1997-04-21 (Actual)

PRIMARY OUTCOMES:
To understand the mechanisms driving eosinophilia and disease pathogenesis in patients with a wide range of eosinophilic disorders | Ongoing assessment
  Identification and characterization of clinical and genetic variants of hypereosinophilic syndromes.

SECONDARY OUTCOMES:
To assess the signs and symptoms experienced by patients with HES | Ongoing
  Creation of a patient-related outcomes questionnaire for use in future treatment studies of HES
To understand the mechanisms of action of therapeutic agents used or in development for the treatment of HES | Ongoing
  Delineation of the effects of therapeutic agents on eosinophil development, activation, recruitment to the tissues and/or apoptosis
To determine the mechanisms underlying eosinophil activation and recruitment to the blood and tissues | Ongoing
  Identification of biomarkers of disease activity and specific organ involvement in eosinophilic disorders; identification of new therapeutic targets for the treatment of HES
To develop a diagnostic algorithm that accurately classifies eosinophilic patients by underlying etiology | Ongoing
  Identification of laboratory and clinical tests that distinguish between clinical and genetic variants

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ezekwe EAD Jr, Khoury P, Nutman TB. Anaphylaxis. J Allergy Clin Immunol Pract. 2024 Jan;12(1):262-263.e12. doi: 10.1016/j.jaip.2023.09.028. No abstract available. PMID 38185496
- [Derived] Stokes K, Yoon P, Makiya M, Gebreegziabher M, Holland-Thomas N, Ware J, Wetzler L, Khoury P, Klion AD. Mechanisms of glucocorticoid resistance in hypereosinophilic syndromes. Clin Exp Allergy. 2019 Dec;49(12):1598-1604. doi: 10.1111/cea.13509. Epub 2019 Oct 27. PMID 31657082
- [Derived] Kuang FL, Legrand F, Makiya M, Ware J, Wetzler L, Brown T, Magee T, Piligian B, Yoon P, Ellis JH, Sun X, Panch SR, Powers A, Alao H, Kumar S, Quezado M, Yan L, Lee N, Kolbeck R, Newbold P, Goldman M, Fay MP, Khoury P, Maric I, Klion AD. Benralizumab for PDGFRA-Negative Hypereosinophilic Syndrome. N Engl J Med. 2019 Apr 4;380(14):1336-1346. doi: 10.1056/NEJMoa1812185. PMID 30943337
- [Derived] Khoury P, Desmond R, Pabon A, Holland-Thomas N, Ware JM, Arthur DC, Kurlander R, Fay MP, Maric I, Klion AD. Clinical features predict responsiveness to imatinib in platelet-derived growth factor receptor-alpha-negative hypereosinophilic syndrome. Allergy. 2016 Jun;71(6):803-10. doi: 10.1111/all.12843. Epub 2016 Mar 2. PMID 26797802
- [Derived] Khoury P, Herold J, Alpaugh A, Dinerman E, Holland-Thomas N, Stoddard J, Gurprasad S, Maric I, Simakova O, Schwartz LB, Fong J, Lee CC, Xi L, Wang Z, Raffeld M, Klion AD. Episodic angioedema with eosinophilia (Gleich syndrome) is a multilineage cell cycling disorder. Haematologica. 2015 Mar;100(3):300-7. doi: 10.3324/haematol.2013.091264. Epub 2014 Dec 19. PMID 25527564
- [Derived] Khoury P, Zagallo P, Talar-Williams C, Santos CS, Dinerman E, Holland NC, Klion AD. Serum biomarkers are similar in Churg-Strauss syndrome and hypereosinophilic syndrome. Allergy. 2012 Sep;67(9):1149-56. doi: 10.1111/j.1398-9995.2012.02873.x. Epub 2012 Jul 9. PMID 22775568
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-I-0079.html